CLINICAL TRIAL: NCT04566068
Title: Adapted Telehealth Intervention for Insomnia Among Cancer Survivors
Brief Title: Survivorship Sleep Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Daniel Hall, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-170
Record Dates: First submitted 2020-09-14; First posted 2020-09-28 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Cancer; Insomnia
Keywords: Insomnia; Cancer Survivors
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention- Adapted Virtual Insomnia Program (Experimental): 4 sessions (approximately 45 min/each, weekly) plus 3 check-ins (approximately 15 min/each, between-sessions) delivered virtually. Sessions are modeled after a published, evidence-based CBT-I protocol and adapted to target needs and preferences identified by cancer survivors. Interventionists will participate in weekly supervision. Approximately half of participants will be asked to wear sleep trackers for one-week prior to starting the intervention (T0) and one-week after completing the intervention (T1).
  Interventions: Behavioral: Intervention- Adapted Virtual Insomnia Program
- Control- Enhanced usual care (Placebo Comparator): Enhanced usual care. Referral to the Massachusetts General Hospital Behavioral Sleep Medicine service plus an educational handout on the topic of sleep hygiene.
  Interventions: Behavioral: Control- Enhanced usual care

INTERVENTIONS:
Behavioral: Intervention- Adapted Virtual Insomnia Program — 4 sessions (approximately 45 min/each, weekly) plus 3 check-ins (approximately 15 min/each, between-sessions) delivered virtually. Sessions are modeled after a published, evidence-based CBT-I protocol and adapted to target needs and preferences identified by cancer survivors.
  Arms: Intervention- Adapted Virtual Insomnia Program
Behavioral: Control- Enhanced usual care — Enhanced usual care. Referral to the Massachusetts General Hospital Behavioral Sleep Medicine service plus an educational handout on the topic of sleep hygiene.
  Arms: Control- Enhanced usual care

SUMMARY:
This is a randomized pilot trial to test the feasibility and acceptability (primary outcomes) of a virtual cognitive behavioral program for insomnia for survivors of various cancer types. Secondary outcomes are to examine the preliminary effects on reducing insomnia severity from baseline to post-intervention.

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy for insomnia (CBT-I), is an evidenced-based insomnia program that is recommended by the American College of Physicians and can be delivered using session-by-session treatment manuals.

Among cancer survivors, CBT-I has only yielded small-to-moderate sized improvements in several aspects of sleep, including sleep efficiency, sleep onset latency, and wake after sleep onset as compared with inactive control conditions. Moreover, systematic reviews of CBT-I with cancer survivors have found high rates of attrition and low attendance. Thus, while CBT-I for cancer survivors is promising, further adaptation is needed to demonstrate greater feasibility and larger effects. Additionally, CBT-I is traditionally delivered in-person, which is not feasible for many cancer survivors. Barriers include time limitations, travel, and illness burden constraints, as well as a paucity of trained CBT-I providers. Telehealth delivery of CBT-I is an innovative approach to address these barriers to care and enhance uptake.

The intervention being tested in this study was informed by a 4-10 session CBT-I protocol and adapted based on interviews the investigators conducted with cancer survivors with insomnia to learn about their sleep-related challenges, suggestions, and preferences for intervention delivery, as well as a systematic review and meta-analysis the investigators published in Sleep Medicine Reviews in 2020.

The research study procedures include screening for eligibility and randomization into 1 of 2 study arms: the Adapted Virtual Intervention Group or a Control Group (Enhanced Usual Care; referral for behavioral sleep medicine and sleep hygiene handout). Participants will be in this research study for approximately 2 months. It is expected that about 40 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* History of nonmetastatic, localized, or regional solid or blood malignancy(ies)
* Completion of primary cancer treatment (i.e., radiation, surgery, and/or chemotherapy)
* Chronic insomnia
* Age ≥18 years

Exclusion Criteria:

* Self-reported inability to speak and write in English
* Undertreated noninsomnia sleep disorder (e.g., sleep apnea)
* Undertreated epilepsy, serious mental illness, or suicidality, and/or psychiatric hospitalization in the past year
* Unwilling or unable to discontinue night shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Feasibility: Enrollment rate of those screened and eligible | T0 (Baseline)- T2(1 Month Post-Intervention Follow Up): 2 Months
  Percent of those screened and eligible who enroll (i.e., sign consent and complete baseline). Reasons for ineligibility, refusal, or drop out, will also be measured along with session attendance.
Acceptability: 5 item measure of enjoyableness, convenience, helpfulness, odds of future use, and overall satisfaction | T0 (Baseline)- T1 (Post-Intervention): 1 Month
  Participants will be asked to rate the enjoyableness, convenience, helpfulness, odds of future use, and overall satisfaction (1=very low to 5=very high) of the program in exit interviews, which will use open-ended questions and response probes to explicate each rating.

SECONDARY OUTCOMES:
Change in Insomnia Severity | T0 (Baseline)- T1(Post-Intervention): 1 Month
  Change in insomnia severity (T0-T1) will be assessed using the validated Insomnia Severity Index (ISI). Scores of 15 or higher on the ISI indicate clinically significant insomnia.

OTHER OUTCOMES:
Exploratory Outcome: Change in nightly subjective sleep and covariance with objective sleep | T0 (Baseline)- T2(1 Month Post-Intervention Follow Up): 2 Months
  Subjective Sleep: Measured via sleep diary (T0-T2). Total sleep time, sleep latency, sleep efficiency, and wake after sleep onset will be assessed using a sleep diary (i.e., timings of sleep/wake, timings of being in bed) for 1-2 weeks to achieve 7 consecutive days of sleep reporting at each timepoint.
Exploratory Outcome: Change in nightly objective sleep and covariance with subjective sleep | T0 (Baseline)- T1(Post-Intervention): 1 Month
  Objective Sleep: Measured via actigraphy data collection (T0-T1). During the same time period as participants complete the sleep diary, objective sleep will be assessed among a subgroup of approximately 10 participants in the intervention arm (counterbalanced) using actigraphy devices to calculate: total sleep time, sleep latency, sleep efficiency, wake after sleep onset, and a Mean Activity Score (actigraph counts/min).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Hall, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Result] Hall DL, Arditte Hall KA, Gorman MJ, Comander A, Goldstein MR, Cunningham TJ, Wieman S, Mizrach HR, Juhel BC, Li R, Markowitz A, Grandner M, Park ER. The Survivorship Sleep Program (SSP): A synchronous, virtual cognitive behavioral therapy for insomnia pilot program among cancer survivors. Cancer. 2022 Apr 1;128(7):1532-1544. doi: 10.1002/cncr.34066. Epub 2021 Dec 16. PMID 34914845
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811